CLINICAL TRIAL: NCT01766349
Title: Effect of Concurrent Chemoradiation Therapy on Respiratory Muscle Performance, Lung Function and Functional Capacity in Patients With Primary Esophagus Cancer
Brief Title: Effect of CCRT on Respiratory Performance and Functional Capacity in Esophagus Cancer Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH-IRB-100066-E
Record Dates: First submitted 2012-12-20; First posted 2013-01-11 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2013-01

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Respiratory muscle strength; Pulmonary function testing; Functional exercise capacity
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- esophagus cancer patients: Respiratory muscle performance will be followed in patients with esophagus cancer during CCRT or RT treatments.
  Interventions: Behavioral: respiratory muscle performance

INTERVENTIONS:
Behavioral: respiratory muscle performance — Respiratory muscle performance will include measurements of respiratory muscle strength and pulmonary function testing.

SUMMARY:
The purposes of this study are to investigate in patients with newly diagnosed esophageal cancer: 1)changes in pulmonary and respiratory muscle function, functional capacity and quality of life during and after RT or CCRT treatment; 2)the correlations between these changes; and 3)the impacts of these changes on the postoperative pulmonary complications following esophagectomy.

DETAILED DESCRIPTION:
Background and Purpose: Incidence rates of esophageal cancer vary internationally with the higher rate found in Eastern Asia. Preoperative concurrent chemoradiation therapy (CCRT) for resectable esophageal cancer has been shown to improve overall survival in meta-analyses. Preoperative pulmonary function and functional capacity are known predictive factors for the development of postoperative pulmonary complications in patient undergoing major cancer surgery. Little is known concerning the impacts of preoperative CCRT on pulmonary function and functional capacity in patients with esophageal cancer. The aim of this study is to examine changes of respiratory performance and functional exercise capacity during RT or CCRT, the relations between these changes, and the impacts of these changes on the postoperative outcomes in patients with esophageal cancer.

Method: Patients with newly diagnosed esophageal cancer without metastasis will be recruited from the Far Eastern Memorial Hospital. Demographic data will be obtained from the chart. Respiratory muscle strength will be measured by maximal inspiratory and expiratory pressure. Spirometric variables will be tested by force expiratory volume in one second and forced vital capacity. Dyspnea will be measured using modified Borg scale. Functional exercise capacity will be measured by six minute walk distance. Quality of life will be measured using EORTC QOL-C30 and QOL-OES18 instruments. All the measurements will be repeated weekly during the concurrent therapy period. Repeated measure ANOVA will be used for analyzing difference among various time points. Spearman correlation coefficient will be used to test relationship between multiple variables. For patients who are receiving esophagectomy after CCRT or RT, pulmonary complications and total length of hospital stay will be documented.

Clinical relevance: The results of this study will help to better understand the indications for chest physiotherapy (e.g., respiratory muscle weakness, reduced functional capacity, and their related sequels)

ELIGIBILITY:
Inclusion Criteria:

* primary esophagus cancer
* planning to receive radiation therapy

Exclusion Criteria:

* MMSE < 24
* A clinical diagnosis affecting respiratory muscle function and functional activity performance
* Unstable angina or acute myocardial infarction prior 1 month of assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with primary esophagus cancer and receive radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes of respiratory muscle performance (MIP/MEP, PFT)from baseline | Baseline, during CCRT or RT treatment (Day 5, Day 10, Day 15, Day 20, Day 25), 2 weeks after the completion of the treatment, 1 day pre-operation, and 1 month after operation
  Maximum inspiratory pressure (MIP) Maximum expiratory pressure (MEP) PFT: FEV1, FVC, FEV1/FVC

SECONDARY OUTCOMES:
Changes of functional exercise capacity, dyspnea, and quality of life from baseline | Baseline, during CCRT or RT treatment (Day 5, Day 10, Day 15, Day 20, Day 25), 2 weeks after the completion of the treatment, 1 day pre-operation, and 1 month after operation
  Functional exercise capacity will be measured using six-minute walk test. Modified Borg scale will be used to measure dyspnea. EORTC QOL-C30 and QOL-OES18 instruments will be used to measure Quality of life.
Prevalence of pulmonary complications | During hospital stay after esophagectomy (average hospitalization after the operation ranges from 1 month to 3 months)
  Data will be retrieved from the chart.
Total length of hospital stay | During hospital stay after esophagectomy (average hospitalization after the operation ranges from 1 month to 3 months)
  Data will be retrieved from the chart.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hsi Hsieh, MD., Ph.D., Principal Investigator — Department of Radiation Oncology, Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial hospital, New Taipei City, Taiwan